CLINICAL TRIAL: NCT07349134
Title: Pilot Randomized Controlled Trial of a Digital Intervention to Promote Wellness, Empowerment, and Lifestyle Learning for Patients With Myeloproliferative Neoplasms (WELL-MPN)
Brief Title: WELL-MPN: A Digital Lifestyle App for Patients With MPNs
Acronym: WELL-MPN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Chi-Joan How, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-805
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Myeloproliferative Neoplasms (MPNs)
Keywords: Myeloproliferative Neoplasms; Essential Thrombocythemia; Polycythemia Vera; Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WELL-MPN Digital App (Experimental): WELL-MPN app and usual care
  Interventions: Behavioral: WELL-MPN Digital App
- Enhanced Usual Care (No Intervention): Usual care and written literature about diet and physical activity guidelines in patients with cancer

INTERVENTIONS:
Behavioral: WELL-MPN Digital App — Patients randomized to the WELL-MPN arm will be given access to the WELL-MPN digital program (app) which provides lifestyle counseling through an iPad.
  Arms: WELL-MPN Digital App

SUMMARY:
The goal of this clinical trial is to learn whether a digital lifestyle app can help improve diet, physical activity, symptoms, emotional well-being, and quality of life in adults with myeloproliferative neoplasms (MPNs).

The main questions it aims to answer are:

Can people with MPNs use the WELL-MPN app?

Does using the WELL-MPN app improve diet quality and physical activity?

Does the WELL-MPN app improve MPN-related symptoms, anxiety and depression, confidence in managing health, and overall quality of life?

Researchers will compare participants who use the WELL-MPN digital app with participants who receive written educational materials about diet and physical activity for people with cancer to see if the app leads to greater improvements in lifestyle behaviors, symptoms, and well-being.

Participants will:

Be randomly assigned to use the WELL-MPN app or receive written lifestyle education materials

Use the assigned program or materials over the study period

Complete surveys about diet, physical activity, symptoms, mood, confidence in self-care, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a myeloproliferative neoplasm (MPN) by World Health Organization 2016 criteria
* Adult (age >/= 18)
* Able to comprehend and speak English
* Able to provide informed consent

Exclusion Criteria:

* Unable to comprehend and speak English
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients consented and enrolled onto the study, and number of patients who complete at least 2 out of 3 modules in the app. | 2 years
  Primary outcome is feasibility, defined as ≥60% enrollment of eligible patients and ≥70% of patients randomized to the intervention group completing at least 2 out of 3 of app modules.
8-Item Client Satisfaction Scores (CSQ-8) | Enrollment to 16 weeks after enrollment
  Acceptability of WELL-MPN as measured by CSQ-8 scores of WELL-MPN. The CSQ-8 is a self-report tool designed to measure patient satisfaction with a received intervention. It consists of 8 items rated on a 4-point Likert scale (from "quite dissatisfied" to "very satisfied"), with higher scores indicating greater satisfaction. WELL-MPN is considered acceptable if >80% of participants on the WELL-MPN arm report a CSQ-8 score >20.

SECONDARY OUTCOMES:
Healthy Eating Index calculated from the Automated Self-Administered Dietary Assessment Tool | Enrollment to 16 weeks after enrollment.
  Diet quality will be compared between control and WELL-MPN patients. The ASA24 is a free 24-hour dietary recall tool developed by the National Cancer Institute. Responses will be used to calculate a Healthy Eating Index (HEI) score, which is a measure of dietary quality that addresses compliance with the 2015 United States Department of Agriculture dietary guidelines (scores range from 0 to 100, with higher scores indicating greater alignment with dietary guidelines).
Mini Eating Assessment Tool (Mini-EAT) score | Enrollment to 16 weeks after enrollment.
  Diet quality will be compared between control and WELL-MPN patients. The Mini-EAT is a 9-item validated brief dietary screener designed for greater ease of administration compared to the ASA-24 but has strong correlation with the HEI. Responses generate a score ranging from 0 to 54, with higher scores reflecting greater adherence to healthy dietary patterns aligned with the Dietary Guidelines for Americans.
Godin Leisure Time Exercise Questionnaire | Enrollment to 16 weeks after enrollment.
  Physical activity will be compared between control and WELL-MPN patients. The Godin Leisure Time Exercise Questionnaire is a brief, self-reported tool used to assess a person's usual physical activity during their free time.It consists of three questions asking information on the number of times one engages in mild, moderate, and strenuous physical activity of at least 15-minute durations in a typical week. Higher scores indicate greater physical activity, with scores of less than 14 units indicating insufficient / sedentary activity.
Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy Short Forms | Enrollment to 16 weeks after enrollment.
  Self-efficacy will be compared between control and WELL-MPN patients. The PROMIS Self-Efficacy Short Forms include 4-item scales across domains such as managing daily activities, symptoms, medications, emotions, and social interactions. Each item is rated on a 5-point Likert scale, with higher scores indicating greater self-efficacy.
MPN Symptom Assessment Form (SAF) Total Symptom Score (TSS) | Enrollment to 16 weeks after enrollment.
  MPN symptom scores will be compared between control and WELL-MPN patients. The MPN SAF TSS is a 10-item questionnaire assessing the most representative and clinically relevant MPN symptoms (concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, fever), and includes a "worst fatigue" question from the Brief Fatigue Inventory. Each subscale ranges from 0 (absent / as good as it can be) to 10 (worst imaginable / as bad as it can be), and scores are computed as the average of the observed items multiplied by 10 to achieve a 0 to 100 scale.
Hospital Anxiety and Depression Scale (HADS-A and HADS-D): | Enrollment to 16 weeks after enrollment.
  Psychological distress will be compared between controls and WELL-MPN patients. The 14-item HADS consists of two 7-item subscales assessing anxiety and depression symptoms in the past week. Each subscale ranges from 0 (no distress) to 21 (maximum distress), with higher scores indicating worse distress. Subscale scores > 8 indicate clinically significant distress; scores can be further interpreted as follows: 8-10 indicates mild distress, 11-14 indicates moderate distress, and 15-21 indicates severe distress.
Functional Assessment of Cancer - General (FACT-G) | Enrollment to 16 weeks after enrollment.
  Quality of life will be compared between controls and WELL-MPN patients. The FACT-G consists of four subscales assessing well-being across four domains (physical, functional, emotional, and social). Subscale scores include Functional Well-Being (0-28), Social Well-Being (0-28), Emotional Well-Being (0-24), and Functional Well-Being (0-28) with higher scores reflecting better well-being in each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Joan How, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States